CLINICAL TRIAL: NCT00829088
Title: An Open Label, Single Dose, Phase I Study of the Excretion of Radioactivity, Metabolism and Pharmacokinetics Following Oral Administration of [14C]AZD2066 to Healthy Male Subjects
Brief Title: Investigation of Rate + Extent of Excretion of Radioactivity in Urine +Faeces After Oral Administration of [14C]AZD2066
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD, PhD, Medical Science Director, Emerging Analgesia, Neuroscience, AstraZeneca R&D Södertälje, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D0475C00008; EudractCT No: 2008-006129-14
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Pain
Keywords: Mass balance; AZD2066; Pain; Pain conditions
MeSH Terms: conditions — Pain | interventions — AZD2066

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD2066 — 1 dose oral solution

SUMMARY:
The aim of this study is to get information about absorption, distribution, metabolism and excretion as well as the tolerability and safety of AZD2066 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Clinically normal physical findings and laboratory values as judged by the investigator and a normal resting ECG.

Exclusion Criteria:

* History of somatic disease/condition, which may interfere with the objectives of the study.
* History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder.
* Healthy volunteers who have been exposed to radiation levels above background (eg, through X-ray examinations).

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Excretion (rate and extent) of radioactivity in urine and faeces following oral administration of [14C]AZD2066 | Until >90% of predicted total radioactivity has been recovered
Pharmacokinetics of total radioactivity in plasma and unchanged AZD2066 in plasma | Sampling at defined timepoints during residential period from pre-dose until 168h post-dose.
Metabolite profile in plasma and excreta | Sampling at defined timepoints during residential period from pre-dose until 48h post-dose.

SECONDARY OUTCOMES:
AZD2066 metabolites in plasma+excreta if feasable | Sampling at defined timepoints during residential period from pre-dose until 48h post-dose.
Safety and tolerability of AZD2066 by assessment of vital signs, laboratory variables, ECG and adverse events | Assessments taken at visit 1 (enrolment), defined time points pre dose and post dose during visit 2 (residential period) and follow up visit 3.

CONTACTS AND LOCATIONS:
Overall Officials: Emeline Ramos, MD, Principal Investigator — AstraZeneca R&D, CPU Alderley Park, UK; Lars Ståhle, MD, Study Chair — AstraZeneca R&D, Södertälje, Sweden
Locations (1):
- Research Site, Cheshire, United Kingdom